CLINICAL TRIAL: NCT05248932
Title: Role of Norepinephrine Infusion in Preventing Hypotension During Spinal Anesthesia for Cesarean Delivery.
Brief Title: Norepinephrine to Prevent Hypotension in Ceasrean Delivery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, mostafa saieed fahim mansour, lecturer, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 19919ANET33
Record Dates: First submitted 2021-12-29; First posted 2022-02-21 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Hypotension; Cesarean Section Complications
Keywords: hypotension; norepinephrine
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- infusion (Active Comparator): patients will receive an infusion of norepinephrine that will be started at 2.5μg/min immediately after intrathecal injection and then manually adjusted according to monitoring of blood pressure (bp), heart rate, fluid responsiveness (thoracic volume variations and stroke volume variations), cardiac index and systemic vascular resistance by using cardiometry, with the objective of maintaining values near baseline
  Interventions: Device: cardiometry; Drug: Norepinephrine infusion
- bolus (Active Comparator): patient with no prophylactic vasopressor and a bolus of 5 μg norepinephrine will be given whenever systolic BP decreases to <80% of the baseline value.
  Interventions: Drug: Norepinephrine bolus; Device: cardiometry

INTERVENTIONS:
Drug: Norepinephrine bolus — 5 microgram bolus therapy
  Arms: bolus
Device: cardiometry — cardiac output, stroke volume and fluid responsiveness monitoring
Drug: Norepinephrine infusion — 2.5 microgram/min infusion
  Arms: infusion

SUMMARY:
This study will be conducted on 40 healthy women having spinal anesthesia for elective cesarean delivery in the operating rooms at Menoufia university hospital.

DETAILED DESCRIPTION:
Informed written consent will be taken from all subjects included in the study after approval of the study by the local ethical committee.

All subjects will be subjected to thorough history taking with risk factors, medical histories, general clinical examination, local clinical examination, laboratory investigations as complete blood count and coagulation profile.

Standardized anesthetic care will be provided according to institutional standards, which include fasting, antacid premedication and noninvasive hemodynamic monitoring After arrival in the operating room, patients will be positioned supine with left lateral tilt, pulse oximeter, ECG leads, non-invasive blood pressure cuff and cardiometry leads (4 surface ECG electrodes is attached to the left side of the neck and the lower thorax (approximately at the level of the xiphoid process) will be attached to patient for monitoring of blood pressure (bp), heart rate, fluid responsiveness (thoracic volume variations and stroke volume variations), cardiac index and systemic vascular resistance and values will be recorded as a baseline and every 10 minutes after intrathecal injection.

10 ml/kg/hr lactated ringer solution will be infused to all patients through an 18 gauge intravenous cannula for 30 minutes as a preload before spinal anesthesia then reduced to maintenance infusion of 6 ml/kg/hr.

Patients will be then placed in sitting position. After skin disinfection and skin infiltration with lidocaine 1%, spinal anesthesia will be performed with 2ml 0.5% hyperbaric bupivacaine (10 mg) in addition to 0.5 ml fentanyl (25 μg) at L3-L4 or L4-L5.

The patient will be then returned to the left-tilted supine position. The study drug regimen will be started immediately after intrathecal injection.

ELIGIBILITY:
Inclusion Criteria:

* ASA I & II
* Non laboring
* Normotensive
* Elective cesarean delivery under spinal anesthesia.
* Baseline systolic blood pressure 90-140 mm Hg

Exclusion Criteria:

* Known fetal abnormality.
* Preexisting or pregnancy-induced hypertension.
* Known cardiovascular or cerebrovascular disease.
* Thrombocytopenia, coagulopathy or any contraindication to spinal anesthesia.
* Weight <50 or >100 kg, height <140 or >180 cm.
* Inability or refusal to give informed consent

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant females
Enrollment: 40 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
throracic volume variations change from baseline | every 10 minutes up to 1 hour
  using cardiometry
cardiac index change from baseline | every 10 minutes up to 1 hour
  using cardiometry
systemic vascular resistance change from baseline | every 10 minutes up to 1 hour
  using cardiometry
stroke volume variation change from baseline | every 10 minutes and up to 1 hour
  using cardiometry

SECONDARY OUTCOMES:
umblical cord gases sample | in the first minute after delivery
APGAR score | after 5 minutes and 10 minutes after delivery
  score from 1 to 10 with the highest score better for neonatal outcome
Non invasive MEAN blood pressure | every 10 minutes and up tp 1 hour
  change from baseline
Heart rate | every 10 minutes and up to 1 hour
  change from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, University Hospitals, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: No